CLINICAL TRIAL: NCT05870501
Title: Synaptic Imaging and Brain Network Activity Following Ketamine in Treatment Resistant Depression
Brief Title: Synaptic Imaging and Network Activity in Treatment Resistant Depression
Acronym: SIGNATURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 297200
Record Dates: First submitted 2023-03-06; First posted 2023-05-23 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2023-09

CONDITIONS: Depressive Disorder; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Bipolar Disorder; Bipolar Disorder I; Bipolar Disorder II; Mood Disorders; Anhedonia
Keywords: Depression; Bipolar Disorder; Major Depressive Disorder; MDD; Treatment-Resistant Depression; Ketamine
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Bipolar Disorder; Mood Disorders; Anhedonia; Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: A double-blind active-placebo crossover design will be used to study a single group of people with TRD to assess the effects of ketamine on brain networks activity versus an active placebo (midazolam). Participants will be randomised to receive three separate IV infusions of ketamine (0.5mg/kg) followed by three separate IV infusions of midazolam (0.045mg/kg), or three separate infusions of midazolam followed by three separate infusions of ketamine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine followed by midazolam (Experimental): Ketamine 0.5mg/kg (three IV infusions) followed by midazolam 0.045mg/kg (three IV infusions)
  Interventions: Drug: Ketamine; Drug: Midazolam
- Midazolam followed by ketamine (Experimental): Midazolam 0.045mg/kg (three IV infusions) follower by ketamine 0.5mg/kg (three IV infusions)
  Interventions: Drug: Ketamine; Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — 0.5mg/kg IV infusion
Drug: Midazolam — 0.045mg/kg IV infusion

SUMMARY:
The main aim of this research is to explore the effects that ketamine has on the functional connectivity of the brain in participants with treatment resistant depression (TRD). This study will investigate the relationship between these changes and response to treatment as measured by clinical scales, as well as examining drug induced changes in reward and emotion based brain activity, structural connectivity, cerebral blood flow, cognition, metabolism and blood markers of brain plasticity.

DETAILED DESCRIPTION:
A double-blind active-placebo crossover design will be used to study a single group of people with TRD to assess the effects of ketamine on brain networks activity versus an active placebo (midazolam). Participants will receive three separate IV infusions of ketamine (0.5mg/kg) followed by three separate IV infusions of an active placebo (midazolam (0.045mg/kg)), or 3 IV infusions of midazolam followed by 3 IV infusions of ketamine. Treatment order will be randomized in a crossover design.

The study will consist of 11 visits including a screening visit, baseline assessments, and two main infusion periods each involving 3 separate IV infusions and a post infusion assessment visit 24 hrs after the third infusion. Ketamine or midazolam will be administered at each of the infusion periods in a crossover design.

Assessment visits will include MRI, EEG and cognitive and clinical assessments.

Up to 50 subjects will be enrolled to ensure that evaluable data is obtained from 45 subjects. The primary comparison will be within-subject between active treatment and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, aged between 18 and 55 years of age inclusive.
* Have a diagnosis of MDD, Bipolar 1 or Bipolar 2 depression and fulfil criteria for TRD depression. TRD patients are defined as having inadequately responded to at least two courses of antidepressants, given in a therapeutic dose and duration (Fekadu et al., 2018).
* Have moderate to severe depression symptoms as demonstrated by a MADRS score greater than 20.
* Be physically healthy, defined as having no clinically relevant abnormalities identified by a detailed medical history and full examination including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests
* Have a good command of the English language.
* Have no or very little knowledge of the Chinese language.
* Provide a personally signed and dated informed consent document indicating that the participant has been informed of and agrees to comply with all aspects of the study.
* Be willing and able to comply with scheduled visits, dosing plan, laboratory trials and any other necessary procedures.

Exclusion Criteria:

* Have a current diagnosed psychiatric disorder, except MDD, Bipolar 1 and Bipolar 2 disorders and comorbid generalised anxiety disorder (GAD), social anxiety and/or social phobia.
* Have a current or previously diagnosed psychotic disorder: Schizophrenia, Schizoaffective Disorder, Delusional disorder, Schizophreniform disorder, Schizotypal (personality) disorder, or Brief psychotic disorder.
* Have previously failed Ketamine as an antidepressant treatment given at a therapeutic dose.
* Have previously experienced an adverse response to ketamine and/or midazolam.
* Have scored 70 or lower in the WASI at the screening visit.
* Have one or more immediate family members with a current or previously diagnosed psychotic disorder.
* Have a medically significant condition which renders them unsuitable for the study (e.g., diabetes, severe cardiovascular disease, severe respiratory disease (e.g. COPD), hepatic or renal failure etc.).
* Be pregnant or breastfeeding, if female.
* Have any MR contra-indications (e.g., metal implants, pacemakers, claustrophobia etc.) which would render them unsuitable for the study.
* Currently consume alcohol in excess of 28 units a week or more than 6 cups of caffeinated drinks per day.
* Smoke more than 5 cigarette per day
* Have taken illicit drugs 7 days prior to admission or current use of drugs of abuse including amphetamines, MDMA, cannabis and opioids Have taken any other medication during the course of the study that has not been discussed. This should be documented by the investigators. (As an exception, 1g paracetamol/24 hours may be taken up to 24 hours prior to any visit).
* Have consumed alcohol or caffeine within 12h and/or nicotine 4h hours prior to the screening visit, study day 1, 2 and 3 and each infusion visit until discharged at the end of each of those visits.
* Have consumed grapefruit juice or Seville oranges-containing products 24 hours prior to admission.
* Have used any prescribed medication in the 3 weeks prior to enrolment or non-prescription medication (other than paracetamol) in the previous 7 days, excluding medication prescribed for bipolar I and II and MDD.
* Have a significant history of drugs of abuse (including benzodiazepines) or positive drugs of abuse test.
* Have received another new chemical entity in the 1 month before dosing or taken part in another research study using drugs within 1 month before dosing.
* Have an acute illness within 2 weeks before the start of study.
* Have any clinically significant abnormalities in clinical chemistry (including liver function tests), haematology or urinalysis results.
* Have self-reported HIV, hepatitis B or hepatitis C
* Have a definite or suspected personal or family history of intolerance or hypersensitivity to drugs and/or their excipients, judged to be clinically relevant by the investigator.
* Have a history or presence of gastrointestinal, hepatic or renal disease or other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Have uncontrolled hypertension, or supine systolic BP outside of the range of 90 to 140 mmHg and a supine diastolic BP outside the range of 40 to 90 mmHg, after a period of acclimatisation.
* Have a decrease in systolic BP of > 25 mmHg or a decrease in diastolic BP of > 15 mmHg when going from resting in bed to standing position, with or without symptoms such as dizziness or light- headedness. (For determination of orthostatic hypotension, lying and standing BP will be recorded after the subject has rested for 10 minutes and has had resting BP recorded followed by measurements 5 minutes after standing)
* Have had treatment in the previous 3 months with any drug known to have a well-defined potential for hepatotoxicity (e.g., halothane).
* Have a risk of suicide according to the investigator's clinical judgment (eg, per C-SSRS positive answer on question 5 within 6 months or has made a suicide attempt within 6 months prior to screening visit).
* Have started a course of hormone replacement therapy within 8 weeks prior to the screening visit.
* Be a subject who, in the opinion of the investigator, should not participate in the study for reasons of safety.
* Have a score of more than 20 on the YMRS at study day 1 and at each subsequent assessment
* Be a subject who, in the opinion of the investigator, has a significant history of mixed episodes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
To investigate the effects of ketamine on brain resting state functional magnetic resonance imaging (fMRI) connectivity in patients with depression compared to placebo | Baseline and 24 hours post third IV infusion
  Change in resting state connectivity measured with fMRI

SECONDARY OUTCOMES:
To investigate the effects of ketamine on fMRI task-based activity during an emotional processing task compared to placebo | Baseline and 24 hours post third IV infusion
  Changes in task related fMRI activity using an emotional processing task (Region of Interest (ROIs): Anterior cingulate cortex (ACC), medial frontal cortex; whole brain analysis)
To investigate the effects of ketamine on fMRI task-based activity during a reward-processing task compared to placebo | Baseline and 24 hours post third IV infusion
  Changes in task related fMRI activity using a reward processing task. (Regions of interest (ROIs): striatal, thalamic and prefrontal regions; whole brain analysis)
To investigate the effects of ketamine on prolactin levels | Baseline and 40 minutes post third IV infusion
  Blood samples analysed for prolactin levels at baseline, pre third infusion and post third infusion of ketamine and placebo
To investigate the effects of ketamine on anhedonic symptoms (as measured by SHAPS) compared to placebo | Baseline and 24 hours post third IV infusion
  The Snaith-Hamilton Pleasure Scale (SHAPS) is a self report scale of hedonic experience and is assessed at baseline and 24 hrs post infusion of ketamine and placebo. The scale ranges from 14-56, with a higher score indicating higher levels of anhedonia
To investigate the effects of ketamine on depression symptoms (as measured by MADRS) compared to placebo | Baseline and 24 hours post third IV infusion
  The Montgomery-Asberg Depression Rating Scale is a interview based scale of depression symptoms and is assessed at baseline of each session and 24 hrs post infusion of ketamine and placebo. The scale ranges from 0-60, with a higher score indicating an higher severity of depression symptoms.
To investigate the effects of ketamine on depression symptoms (as measured by QIDS) compared to placebo | Baseline, pre infusion and 24 hours post third IV infusion
  The Quick Inventory of Depressive Symptomatology-Self Report (QIDS) is a self report scale of depression symptoms and is assessed at baseline, pre infusion and 24 hrs post third infusion of ketamine and placebo The scale ranges from 0-42, with a higher score indicating an higher severity of depression symptoms.
To investigate the effects of ketamine on the M3VAS compared to placebo | Baseline, pre infusion and 24 hours post third IV infusion
  The Maudsley 3-item Visual Analogue Scale (M3VAS) is a self report visual analogue scale (VAS) of three main domains of depression symptoms (mood, pleasure and suicidality) and is assessed at baseline, pre infusion and 24 hrs post third infusion of ketamine and placebo. The VAS ranges from 0-100 on each domain, with a higher score indicating an higher severity of that domain.
To investigate the effects of ketamine on brain perfusion (ASL) compared to placebo | Baseline and 24 hours post third IV infusion
  Arterial spin labelling (ASL) is a measure of blood flow or perfusion in the brain. Measures are taken at baseline and 24 hours post third infusion of ketamine and placebo
To investigate the blood plasma concentration (μg/mL) of ketamine following the third IV infusion | 40 minutes, 120 minutes, 200 minutes and 24 hours post third IV infusion
  Blood samples will be taken to measure the blood concentration of ketamine at specific time points post infusion
To investigate the blood plasma concentration (μg/mL) of hydroxynorketamine following the third IV infusion | 40 minutes, 120 minutes, 200 minutes and 24 hours post third IV infusion
  Blood samples will be taken to measure the blood concentration of hydroxynorketamine (a metabolite of ketamine) at specific time points post infusion
To investigate the blood plasma concentration (μg/mL) of norketamine following the third IV infusion | 40 minutes, 120 minutes, 200 minutes and 24 hours post third IV infusion
  Blood samples will be taken to measure the blood concentration of norketamine (a metabolite of ketamine) at specific time points post infusion
To investigate the effects of ketamine on a short battery of cognitive tasks compared to placebo | Baseline 24 hours post third IV infusion
  The Cognition is a self administered web-based battery of cognitive tasks that will be conducted at baseline, and 24 hours post third infusion of ketamine and placebo
To investigate the effects of ketamine on blood biomarkers related to synaptogenesis compared to placebo | Baseline and 24 hours post third IV infusion
  Blood samples taken at baseline and 24 hours post third infusion of ketamine and placebo will be analysed for markers of synaptic plasticity (Brain derived neurotrophic factor (BDNF))
To investigate the effects of ketamine on the power of frequency bands (alpha, theta, gamma) in resting EEG | Baseline and 24 hours post third IV infusion
  Electroencephalogram (EEG) is an brain imaging technique that allows the recording of brain electrical activity and will be conducted at baseline, and 24 hours post third infusion of ketamine and placebo
To investigate the effects of ketamine on structural connectivity (DTI) compared to placebo | Baseline and 24 hours post third IV infusion
  Diffusion tensor imaging (DTI) is a measure of brain tissue microstructure. Measures are taken at baseline and 24 hours post third infusion of ketamine and placebo
To investigate the effects of ketamine on visual and auditory based ERPs compared to placebo | Baseline and 24 hours post third IV infusion
  Event related potentials (ERPs) are an EEG measure related to brain electrical activity that can be produced by visual and auditory stimuli

OTHER OUTCOMES:
To investigate the effects of ketamine on the cerebral metabolic rate of oxygen utilization (CMRO2) as a measure of brain tissue metabolism using fMRI | 24 hours post third IV infusion
  The cerebral metabolic rate of oxygen can be assessed using specialised fMRI pulse sequences
Baseline measures of common genetic markers (SNPs) for genetic disease risk load | Baseline measure
  Blood samples taken at baseline will be used for DNA analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mitul Mehta, PhD, Principal Investigator — King's College London
Locations (1):
- The Institute of Psychiatry, Psychology & Neuroscience, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT05870501/ICF_000.pdf